CLINICAL TRIAL: NCT03888586
Title: Comparison of Dry Needling and Deep Friction Massage in Patients With Subacromial Pain Syndrome: 1-year Follow-up of a Randomized Controlled Trial
Brief Title: Comparison of Dry Needling and Deep Friction Massage in Patients With Subacromial Pain Syndrome
Acronym: Dry Needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Başar Öztürk, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: manualpt2019
Record Dates: First submitted 2019-03-22; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Subacromial Impingement Syndrome; Trigger Point Pain, Myofascial
Keywords: Dry needling, subacromial joint, night pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Experimental): Participants were administered trigger point dry kneedling technique 6 times for 1 month, once every 5 days. The subject was positioned prone and the arm position was slightly changed related with the muscle. After the skin inspection it was cleaned with the alcohol. .
  Interventions: Device: Trigger Point Dry Needling Technique
- Deep Friction Massage (Experimental): Deep friction massage was applied transversely unlike the superficial massage and sufﬁciently deep to the ﬁber direction of affected connective tissue to maintain the mobility. Totally 6 sessions were administered twice a week for 3 weeks.
  Interventions: Other: Deep Friction Massage Technique

INTERVENTIONS:
Device: Trigger Point Dry Needling Technique — The type of needle and the depth of the entrance varied depending on the estimated muscle thickness (0.25 - 25 mm, 0.25 - 30 mm and 0.25-40 mm). The disposable stainless-steel sterile needles were inserted through the skin over the trigger point in the taut band of muscle using the fast-in/out technique. Forward and backward needling was repeated until the local twitch responses were obtained. The depth of the needle was changed depending on the muscle thickness. After the first local twitch response, the needle was moved up and down 3 to 5 mm in only vertical directions until no more local twitch responses were elicited. After removing the needle, the insertion area was compressed with a piece of cotton
  Arms: Dry Needling
Other: Deep Friction Massage Technique — For supporting the normal healing conditions, the deep and transverse friction causes hyperaemia in the involved soft tissue, which results in increased blood ﬂow to the area.
  Arms: Deep Friction Massage

SUMMARY:
This study was planned to investigate the effects of Trigger Point-Dry Needling Therapy (TP-DNT) on night pain and Shoulder Internal Rotation (SIR) in individuals with Subacromial Pain Syndrome (SPS).

DETAILED DESCRIPTION:
Shoulder pain seen intensely in the general population, many methods has been used for the treatment which has not been fully proven to be superior to each other. Before considering surgical approaches, trying conservative approaches is emphasized. While literature showed us that nighttime pain is an important musculoskeletal symptom, may be associated with local inflammation, it is an important feature during the treatment planning. TP-DNT had positive effects on night pain and SIR in SPS. It was seen that the treatment satisfaction level of participants was high. Despite these positive findings, there is need for further studies in which sample size is increased, control group is added, and long-term follow-up is planned.

ELIGIBILITY:
Inclusion Criteria:

* To be able to read and speak Turkish well enough to give informed consent and follow the working instructions.
* Having complaints of unilateral shoulder pain for at least 6 months and being diagnosed with subacromial impingement syndrome.
* Having night pain
* Having active trigger point.

Exclusion Criteria:

* Bilateral shoulder pain
* If there is a contraindicated condition for needles such as fear of needles or infection
* History of bleeding disorder
* Shoulder fracture and / or dislocation history
* Symptoms of cervical radiculopathy and / or neuropathy
* The use of antiaggregants, anticoagulants, analgesics or antiinflammatory drugs or drug-like substances (1 week before or during treatment)
* Fibromyalgia syndrome
* Any neurological, motor, or sensory disorder in the upper extremity
* History of surgery on shoulder or neck
* Conservative or invasive physical therapy or infiltration for the shoulder region during the last 6 months
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-02-11 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 1 month
  The VAS was used to measure the mean pain intensity of rest time activity and night time over the previous 3 days . The 10-cm scale was marked with "0" (no pain) and "10" (worst imaginable pain), and the patients were instructed on how to use the scale.

SECONDARY OUTCOMES:
Range of Motion | 1 month
  The goniometric measurement method measures the range of active internal movements of the internal rotation with pre-treatment and after 8 sessions. The movement is repeated 3 times and recorded with the average.
Shoulder Pain and Disability Index (SPADI) | 1 month
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain.
Hospital Anxiety and Depression Scale (HADS) | 1 month
  The HADS aims to measure symptoms of anxiety and depression and consists of 14 items, seven items for the anxiety subscale (HADS Anxiety) and seven for the depression subscale (HADS Depression). HADS Anxiety focus mainly on symptoms of generalized anxiety disorder and HADS Depression is focused on anhedonia, the main symptom of depression. Each item is scored on a response-scale with four alternatives ranging between 0 and 3. After adjusting for six items that are reversed scored, all responses are summed to obtain the two subscales.
Nothingham Health Profile | 1 month
  NHP is a general quality-of-life questionnaire that measures health problems that a person perceives and how these problems affect normal daily activities. The questionnaire consists of 38 items and evaluates six dimensions of health status: energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items) and physical activity (8 matter). Questions are answered yes or no. Each section is scored from 0 to 100 points. 0 indicates the best health status, 100 worst health status. NHP score and total NHP score were evaluated. Total NHP score was obtained from the sum of the sub-scores

CONTACTS AND LOCATIONS:
Locations (1):
- Başar Öztürk, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided